CLINICAL TRIAL: NCT03351452
Title: Effects of Transcranial Electric Stimulation on Associative Memory Formation in Healthy Elderly Participants as Well as in Individuals With Memory Impairment
Brief Title: tES Effects on Associative Memory Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-01197
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real tDCS (Experimental): 20 min of 2 mA real anodal transcranial direct current stimulation applied via 5x7 cm rubber electrode over the VLPFC (current density: 0.057 mA/cm2) and cathodal 10x10 rubber electrode over supraorbital region (current density: 0.02 mA/cm2). Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real anodal transcranial direct current stimulation
- Real tACS (Experimental): 20 min of 2 mA real transcranial alternating current stimulation in theta frequency applied via 5x7 cm and 10x10 cm rubber electrodes over the VLPFC (current density: 0.057 mA/cm2) and supraorbital region (current density: 0.02 mA/cm2). Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real transcranial alternating current stimulation
- Sham tES (Sham Comparator): 30 s of 2 mA sham transcranial electric current stimulation applied via 5x7 cm and 10x10 cm rubber electrodes over the VLPFC (current density: 0.057 mA/cm2) and supraorbital region (current density: 0.02 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the encoding phase of the memory task.
  Interventions: Device: sham transcranial electric current stimulation

INTERVENTIONS:
Device: real anodal transcranial direct current stimulation — The MR-compatible neuroConn DC-Stimulator MR (neuroCare Group, Ilmenau, Germany) will be used.
  Arms: Real tDCS
Device: real transcranial alternating current stimulation — The MR-compatible neuroConn DC-Stimulator MR (neuroCare Group, Ilmenau, Germany) will be used.
  Arms: Real tACS
Device: sham transcranial electric current stimulation — The MR-compatible neuroConn DC-Stimulator MR (neuroCare Group, Ilmenau, Germany) will be used.
  Arms: Sham tES

SUMMARY:
Previous studies showed that transcranial electric stimulation (tES) applied over the prefrontal cortex improves cognitive performance in healthy elderly adults as well as in patients suffering from mild cognitive impairment or early Alzheimer's disease. Therefore, tES methods might be a useful intervention tool for patients suffering from memory impairment in early terms of the disease.

The present study aims at establishing a connection between the stimulation-induced changes on associative memory performance and its underlying neurophysiological parameters. tES effects and their underlying mechanisms will be compared between healthy elderly controls and clinical study populations receiving either real or sham tES over the left ventrolateral prefrontal cortex during an associative memory task.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Non-smokers
* Right-handedness
* Native German speakers or comparable level of fluency
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Neurological or psychiatric condition (other than diagnosed cognitive impairment)
* Past head injuries
* Magnetizable implants
* History of seizures
* Current or life-time alcohol or drug abuse
* Skin diseases

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Performance on immediate cued recall task | 20 min
  Number of correct responses on retrieval task of previously learned associative memory items
Performance on delayed cued recall task | 24 hours
  Number of correct responses on retrieval task of previously learned associative memory items

SECONDARY OUTCOMES:
task-dependent BOLD activity | 20 min
  Measured with functional magnetic resonance imaging (fMRI)
resting-state BOLD activity | 10 min
  Measured with functional magnetic resonance imaging (fMRI)

OTHER OUTCOMES:
Performance on cued recall task | follow-up after 24 hours
  Number of correct responses on retrieval task of previously learned associative memory items
Performance on recognition task | follow-up after 24 hours
  Number of correct responses on retrieval task of previously learned associative memory items

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof.Dr.med, Principal Investigator — University of Bern
Locations (1):
- University Hospital of Old Age Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No